CLINICAL TRIAL: NCT02403661
Title: The Effectiveness of a New Treatment for Patients With Peripheral Nerve Injuries in the Upper Limb
Brief Title: Electrical Stimulation to Enhance Peripheral Nerve Regeneration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00000973
Record Dates: First submitted 2015-03-16; First posted 2015-03-31 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post surgical electrical stimulation (Active Comparator): Balanced AC pulse at 20 Hz with less than 30V and 0.01 ms duration will be delivered for 1 hour.
  Interventions: Procedure: Post surgical electrical stimulation
- Sham stimulation (Placebo Comparator): Stimulation with the same parameters delivered only for 5 s.
  Interventions: Procedure: Post surgical electrical stimulation

INTERVENTIONS:
Procedure: Post surgical electrical stimulation — Post surgical electrical stimulation immediately after surgical nerve repair
  Other Names: electrical stimulation

SUMMARY:
The primary goal of this study is to quantify the functional deficits caused by injuries to the brachial plexus and peripheral nerve in the arm. The second goal is to test the possible benefit of electrical stimulation of the injured nerve following surgery. The investigators will test whether electrical stimulation will improve hand function and nerve regeneration after repair for nerve injury. Injuries causing nerve damage in the arm and hand are common. In severe cases, functional outcomes even with surgery remain poor. Recently, electrical stimulation has been applied to injured nerves in rats. This was shown to improve nerve regeneration. These studies showed that as little as one hour of electrical stimulation was effective. Therefore, the investigators plan to test this new method of treatment to determine whether it is also helpful in humans. These will be done by using a symptom severity questionnaire, nerve conduction studies and by testing pressure sensations, hand dexterity and strength. The patients will be randomized to either the treatment or control group. Following the treatment, all baseline measurements will be reevaluated every three months for the first year and every 6 months during the second year. The timing and nature of the evaluation process will be identical in both groups.

DETAILED DESCRIPTION:
Background Rationale:

Surgical repair and nerve grafting are currently the standard treatment for nerve laceration. However, even with that, the functional outcome in patients with proximal nerve cut is often poor. In those cases, the surviving axons in the proximal nerve stump have already reached their capacity limit to sprout and to reinnervate. Therefore, no further reinnervation can occur even with surgery unless regeneration and extension of the proximal stump can somehow be enhanced. Unfortunately, although many attempts, none were shown to be effective in the clinical setting.

Post-surgical electrical stimulation:

Recent studies demonstrated that electrical stimulation applied directly to an injured peripheral nerve resulted in marked improvement of nerve regeneration. Preliminary data suggesting that electrical nerve stimulation could possibly enhance nerve regeneration has in fact been known for some time. Accelerated rate of regeneration was found in animals that received electrical stimulation for as little as 1 hour. Furthermore, preferential growth of the regenerating sensory axons into the appropriate nerve branch was also accelerated with electrical stimulation.

Since these studies showed that as little as one hour of electrical stimulation was effective in accelerating nerve regeneration, it opens the possibility of applying this to humans. The intervention is safe and of minimal discomfort. Furthermore, the use of electrical stimulation as a clinical treatment modality is already well accepted. In a recent study, the investigators applied this to patients with severe median nerve compressive injury in the carpal tunnel following surgery. The procedure was well tolerated with no adverse event observed in any of the 21 subjects after 1 year of follow up. In fact, compared to the control subjects who received surgery alone, those in the treatment groups showed quicker resolution of their symptoms and more vigorous motor nerve regeneration.

The problem of prolonged denervation:

Prognosis following severe trauma to nerves in the upper arm and forearm, if left untreated, is extremely poor. Current conventional treatment is through primary nerve repair and by inserting a nerve graft (most commonly using the sural nerve) to restore nerve continuity. However, even with that, the extent of reinnervation is often far from complete. The glacial rate of nerve regeneration, at no more than 1 mm a day, can easily leave the target intrinsic hand muscles deprived of nerve innervation for a year or more. The long period of denervation, coupled with a lack of active movements can lead a whole host of negative consequences including muscle fibre fibrosis, contracture, secondary joint derangement and not infrequently, pain. Equally important is the Schwann cells' ability to support trophic support and nerve growth guidance also gradually declines. Therefore, a more effective treatment is urgently needed. A recent approach is by doing a distal nerve transfers. That shortens the distance of reinnervation greatly. However, the outcome following this transfer or with primary suture repair following acute median or ulnar nerve laceration is relatively poor. Another closely related common trauma to the hand is laceration of digital nerves where recovery of sensory functions following primary nerve suture is equally poor. To potentially further expedite the reinnervation, the investigators proposed to additionally stimulate the proximal nerve stump immediately following the nerve transfer and/or the nerve repair. Whether this novel approach will indeed further expedite the reinnervation and improve hand function following nerve laceration is not known at this point. This will be the first human application study to address that question.

Hypothesis/Research Question/Objectives:

Investigators hypothesize that nerve regeneration in the nerves in the arm and digital nerve in the hand can be significantly enhanced when they are combined with post-surgical electrical stimulation. Furthermore, the improved nerve regeneration with post-operative electrical stimulation will result in a significant improvement in hand functions compared with surgery alone.To test these hypotheses, the objectives of this study are to: 1) quantify the functional and physiological consequence of severe nerve injury in the arm, and 2) to compare the outcome of conventional nerve surgery alone versus nerve surgery followed by post-operative electrical stimulation.

Basic Study Design:

Subjects Patients with severe trauma to the nerves in the upper limb resulting in complete axonal loss will be recruited. These patients will be randomly assigned to either nerve repair/transfer alone or nerve repair/transfer followed by one hour of low frequency electrical stimulation. The patients will be followed at 3 month intervals for 2 years.

Post-surgical outcome including electrophysiological evaluation will be done by an independent physician who is not part of the investigation team. Therefore, the testers will not be aware of whether the subjects are in the conventional surgery group or in the surgery+electrical stimulation group.

Interventions

Once all the baseline studies have been completed, the subject will be randomized to one of two groups:

i) Surgery followed by sham stimulation for 5 seconds. Nerve repair/transfer surgery will be performed by a peripheral nerve surgeon.

ii) Surgery followed by 1 hour of electrical stimulation. Electrical stimulation will be done by inserting a pair of fine wires insulated all around except over the most distal 1 cm at the tip through the incision site. Tips of the fine wires will be seated over the proximal nerve stump to depolarize the axons. These fine wire electrodes will be connected to a portable electrical stimulator (model SD9, Grass Instruments, Providence, RI, USA). Continuous 20 Hz electrical stimuli will be delivered at an intensity of 1.5 times of motor threshold for an hour. At this low intensity, there should be little if any discomfort with the stimulation procedure. In a previous series of carpal tunnel syndrome patients carried out at University of Alberta, this was found to be totally safe and well tolerated. The fine wires will be removed once the stimulation protocol is completed.

Methods of outcome evaluation

1. Sensory nerve conduction study to measure the sensory nerve action potential amplitudes.
2. Motor nerve conduction study to measure the compound muscle action potential amplitudes.
3. Motor unit number estimate. The 'multiple point stimulation' technique will be used.
4. Light touch and pressure sensation. This will be tested using the Semmes-Weinstein Monofilaments and McKinnon-Dellon Disk-Criminator.
5. Hand function tests. This will be tested using Moberg Pick-Up Test, Purdue Pegboard Test, Jamar dynamometer for grip strength, Pinch dynamometer for key, tripod and tip-to-tip strength.

Post intervention evaluations:

Following the intervention, all the baseline parameters will be reevaluated every 3 to 6 months for 2 years. The timing and nature of the evaluation procedure will be identical in all the patients.

Statistical Considerations in the study design Since this will be the first human application study for nerve laceration on a novel technique, its results will be valuable in guiding future full scale studies. The rationale for proposing a total 80 subjects in this study is based on a recently completed study on using post surgical electrical stimulation to enhance nerve regeneration in patients with carpal tunnel syndrome. In that randomized controlled study, a similar sample size was used and the investigators found a significant improvement in nerve regeneration in the treatment group compared to controls. Based on motor unit number estimation, the primary outcome used, the treatment group showed a statistically significant improvement compared to the control group.

Data Analysis:

Statistical analysis of changes in the outcome measure parameters within each subject will be done using paired t-test. A p <0.05 will be considered significant. Differences in treatment outcome between the two groups will be done using independent t-test with the treatment method being the independent variable.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe injury to the brachial plexus causing complete denervation.

Exclusion Criteria:

* The presence of other neurologic conditions.
* Cognitive compromise that renders the patients unable to understand and consent to the study.
* Minors younger than the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-03; Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in the sensory nerve action potential amplitude (uV) at 2 years . | preop, every 3 to 6 months for 2 years

SECONDARY OUTCOMES:
Change in the compound muscle action potential amplitude (mV) at 2 years | preop, every 3 to 6 months for 2 years
Change in the motor unit number estimation at 2 years | preop, every 3 to 6 months for 2 years
Change in the ability to perform hand function at 2 years. | preop, every 3 to 6 months for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ming Chan, MB ChB, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Gordon T, Amirjani N, Edwards DC, Chan KM. Brief post-surgical electrical stimulation accelerates axon regeneration and muscle reinnervation without affecting the functional measures in carpal tunnel syndrome patients. Exp Neurol. 2010 May;223(1):192-202. doi: 10.1016/j.expneurol.2009.09.020. Epub 2009 Oct 1. PMID 19800329
- [Result] Al-Majed AA, Tam SL, Gordon T. Electrical stimulation accelerates and enhances expression of regeneration-associated genes in regenerating rat femoral motoneurons. Cell Mol Neurobiol. 2004 Jun;24(3):379-402. doi: 10.1023/b:cemn.0000022770.66463.f7. PMID 15206821
- [Result] Brushart TM, Jari R, Verge V, Rohde C, Gordon T. Electrical stimulation restores the specificity of sensory axon regeneration. Exp Neurol. 2005 Jul;194(1):221-9. doi: 10.1016/j.expneurol.2005.02.007. PMID 15899259